CLINICAL TRIAL: NCT06957743
Title: Mechanisms of Mindfulness Meditation and Self-Hypnosis for Pain in Older Adults With Chronic Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: The University of Queensland (Other); University of Florida (Other); University of California, San Diego (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mark Jensen, Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00021167; R01AG079832-01 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-05-04 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; Mindfulness Meditation; Self-Hypnosis
Keywords: Chronic Pain; Mindfulness Meditation; Self-Hypnosis
MeSH Terms: conditions — Chronic Pain | interventions — Mindfulness; Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mindfulness Meditation (Experimental): Participants will lie flat on their back with their eyes closed and will listen to the clinician read a standardized Mindfulness Meditation script.
  Interventions: Behavioral: Mindfulness Meditation
- Self-Hypnosis (Experimental): Participants will lie flat on their back with their eyes closed and will listen to the clinician read a standardized hypnotic script.
  Interventions: Behavioral: Self-Hypnosis
- Attention Control Condition (No Intervention): Participants in the control condition will listen to four, 20-min. excerpts from a natural history book. The sessions will be done in the same setting as the Mindfulness Meditation and Self-Hypnosis sessions; control participants will lie flat on their back and will listen to the clinician read the standardized book excerpt. This control was chosen as past research has found that individuals who listen to this standardized text report it to be a neutral, but relaxing text, and it has been used as an effective control compared with meditation conditions in previous research.

INTERVENTIONS:
Behavioral: Mindfulness Meditation — The Mindfulness Meditation trainings will teach participants Shamatha Vipassana, which is the specific form of Mindfulness Meditation typically implemented in mindfulness research. The emphasis is placed upon developing focused attention on an object of awareness, such as the breath. This focus is then expanded to include a more open, non-judgmental monitoring of any sensory, emotional, or cognitive events. Participants will be invited to lie flat on their back (i.e., to mimic conditions in the MRI scanner) and will listen to the clinician read a standardized Mindfulness Meditation script.
  Arms: Mindfulness Meditation
Behavioral: Self-Hypnosis — In the Self-Hypnosis group, participants will relax with their eyes closed and, as with Mindfulness Meditation, will lie flat on their lack and will listen to the clinician read a standardized hypnotic script. The Self-Hypnosis practice will include an induction followed by suggestions for decreased pain and improvement in comorbid symptoms (e.g., mood).
  Arms: Self-Hypnosis

SUMMARY:
The goal of this study is to better understand how two common psychological treatments for pain work in the brain of older adults living with chronic pain. This study will:

1. evaluate fMRI of adults receiving psychological treatments for chronic pain relative to an attention control condition to determine how these interventions work within older adults, and
2. examine self-report and EEG variables to identify for whom do these psychological interventions work.

Adults ages 60 years and older, living with chronic pain for at least 3 months will be randomly assigned to one of three conditions:

1. Mindfulness-Meditation
2. Self-Hypnosis
3. Audio Recording Control

DETAILED DESCRIPTION:
Research has shown that psychological treatments can help people with chronic pain manage their pain and improve their quality of life. Two common psychological treatments for chronic pain include Mindfulness-Meditation and Self-Hypnosis. While research has shown these treatments are helpful for people with chronic pain, the benefits people experience from these types of treatments can vary from person to person. There is little research showing who responds best to which treatments and what happens in the brain during these treatments to reduce pain. The purpose of this study is to better understand how these pain treatments work in the brain. By identifying how these pain treatments work to help reduce chronic pain, the study investigators aim to improve treatments for people with chronic pain in the future.

Participants will be asked to attend 7 sessions and complete assessments in-person and online. Study sessions will consist of EEG assessment (in-person session 1), self-report measures (mixed in-person and online, all sessions), MRI and fMRI with concurrent experimental pain stimulation via heat and mechanical pain induction (in-person sessions 2 and 7) and Mindfulness-Meditation or Self-Hypnosis practice (in-person session 7 only), as well as training in Mindfulness-Meditation, Self-Hypnosis, or audio recording control (online sessions 3-6). Participants will spend about 6.5 hours in this study over a 3-week period.

ELIGIBILITY:
Inclusion Criteria:

1. be ≥60 years of age;
2. have self-reported chronic pain (≥3-months, with pain experienced on ≥ 50% of days);
3. endorse an average intensity of pain ≥3 on a 0-10 numerical rating scale (NRS) for most days of the previous 3-months;
4. be able to read, speak, and understand English;
5. be naïve to meditation and hypnosis (<20-min. practice/week over the past 6-months; never attended a mindfulness or self-hypnosis course); and
6. if currently taking analgesic or psychotropic medication, medication must have been stabilized for ≥4-weeks prior to this study.

Exclusion Criteria:

1. have a history of a medical condition that could produce an abnormal EEG (e.g., epilepsy, history of traumatic brain injury);
2. have metals in the body (e.g., clips, prosthetics, pace-makers);
3. self-report claustrophobia or other contraindications to MRI scanning;
4. have uncontrolled hypertension;
5. have a primary chronic pain condition of headache;
6. show signs of cognitive impairment (6-Item Cognitive Screener during screening; MoCA score at Session 1, using demographically-adjusted normative cut-offs that take into account race, ethnicity, and age);
7. have chronic pain due to malignancy (e.g., cancer) or a chronic pain condition for which surgery is recommended and/or planned;
8. are currently receiving other psychosocial treatments for any pain condition (as this may influence these treatment results);
9. self-report previous participation in an experimental pain study; or
10. report <2 on a 0-10 NRS for pain intensity in response to experimental "heat" pain stimuli (in order to avoid floor effects and to ensure participants are not too insensitive to thermal pain to reliably produce detectable pain-related brain activation).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in average chronic pain intensity in past 24 hours | Collected daily for 4 consecutive days at pre-baseline, once at 1-week post-baseline MRI/fMRI assessment, and daily for 4 consecutive days starting day 11 post-baseline MRI/fMRI assessment
  Change in average chronic pain intensity in the past 24 hours will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their chronic pain intensity in the past 24 hours. Higher scores indicate higher levels of self-reported pain intensity. The four daily assessments will be averaged and change scores will be calculated between pre- and post-treatment.

SECONDARY OUTCOMES:
Change in pain threshold | Collected during EEG procedure, baseline MRI/fMRI assessment, and 1-week post-baseline MRI/fMRI assessment
  Change in pain threshold will be measured by noting the point at which the stimulus (temperature/pressure) is detected as 'painful'.
Change in pain tolerance | Collected during EEG procedure, baseline MRI/fMRI assessment, and 1-week post-baseline MRI/fMRI assessment
  Change in pain tolerance will be measured by noting the point at which the stimulus (temperature/pressure) is discontinued.
Change in peak experiment-induced pain intensity | Collected during EEG procedure, baseline MRI/fMRI assessment, and 1-week post-baseline MRI/fMRI assessment
  Change in pain intensity will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their current pain intensity as assessed during the pain stimulus session; the question is asked at the point that pain tolerance is reached. Higher scores indicate higher levels of self-reported pain intensity.
Change in peak experiment-induced pain unpleasantness | Collected during EEG assessment visit, baseline MRI/fMRI assessment, and 1-week post-baseline MRI/fMRI assessment
  Change in pain unpleasantness will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their current pain unpleasantness as assessed during the pain stimulus session; the question is asked at the point that pain tolerance is reached. Higher scores indicate higher levels of self-reported pain unpleasantness.
Change in current pain intensity | Collected during EEG procedure, baseline MRI/fMRI assessment, at each of the 4 treatment sessions, and at 1-week post-baseline MRI/fMRI assessment
  Change in current pain intensity will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their current pain intensity. Higher scores indicate higher levels of self-reported pain intensity.
Change in current pain unpleasantness | Collected during EEG assessment visit, baseline MRI/fMRI assessment, at each of the 4 treatment sessions, and at 1-week post-baseline MRI/fMRI assessment
  Change in current pain unpleasantness will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their current pain unpleasantness. Higher scores indicate higher levels of self-reported pain unpleasantness.
Change in average chronic pain unpleasantness in past 24 hours | Collected daily for 4 consecutive days at pre-baseline, and daily for 4 consecutive days starting day 11 post-baseline MRI/fMRI assessment
  Change in average chronic pain unpleasantness in the past 24 hours will be measured using a 0-10 numerical rating scale. Participants will be asked to choose a number from 0-10 that best represents their chronic pain unpleasantness in the past 24 hours. Higher scores indicate higher levels of self-reported pain unpleasantness.
Change in pain interference | Collected once at pre-baseline, and once on day 13 post-baseline MRI/fMRI assessment
  Change in pain interference with different activities/aspects of life will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4-item short form. Responses from each item will be summed for a total raw score from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported pain interference with different activities/aspects of life.
Change in sleep disturbance | Collected once at pre-baseline, and once on day 13 post-baseline MRI/fMRI assessment
  Change in sleep disturbance will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance 4-item short form. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate more self-reported sleep disturbance.
Change in depression | Collected once at pre-baseline, and once on day 13 post-baseline MRI/fMRI assessment
  Change in depression will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 4-item short form. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher self-reported levels of depression.
Change in fatigue | Collected once at pre-baseline, and once on day 13 post-baseline MRI/fMRI assessment
  Change in fatigue will be measured with the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue 4-item short form. Responses from each item will be summed to form a total raw score ranging from 4-20. The raw scores are then converted to T-Scores, with a mean of 50 and a SD of 10. Higher scores indicate higher self-reported levels of fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jensen, PhD, Principal Investigator — University of Washington; Melissa Day, PhD, Principal Investigator — The University of Queensland

IPD SHARING:
Plan to Share IPD: Yes
The self-report data and metadata will be archived in the Mendeley Data generalist repository. The EEG and fMRI data will be archived in the NeuroImaging Tools & Resources Collaboratory Image Repository (NTRC-IR), which is a NIH-sponsored repository for neuroimaging data.
Supporting Information: Study Protocol
Time Frame: All data will be archived by the time that the award ends. The data will be preserved in the repositories for as long as those repositories continue to exist and curate the data.
Access Criteria: At two years after the end of the project period or after the primary study papers have been published, whichever comes first, access to the data will be granted following completion of a data management and sharing plan agreement with the Department of Rehabilitation Medicine at the University of Washington. Two years after the end of the project period or after the primary study papers have been published, all of the study data will be available to scientists without these scientists needing to complete and sign the UW Department of Rehabilitation's data sharing plan agreement.

REFERENCES:
- [Background] Jensen MP, Patterson DR. Hypnotic approaches for chronic pain management: clinical implications of recent research findings. Am Psychol. 2014 Feb-Mar;69(2):167-77. doi: 10.1037/a0035644. PMID 24547802
- [Background] Patterson DR, Jensen MP. Hypnosis and clinical pain. Psychol Bull. 2003 Jul;129(4):495-521. doi: 10.1037/0033-2909.129.4.495. PMID 12848218
- [Background] Jensen MP, Mendoza ME, Ehde DM, Patterson DR, Molton IR, Dillworth TM, Gertz KJ, Chan J, Hakimian S, Battalio SL, Ciol MA. Effects of hypnosis, cognitive therapy, hypnotic cognitive therapy, and pain education in adults with chronic pain: a randomized clinical trial. Pain. 2020 Oct;161(10):2284-2298. doi: 10.1097/j.pain.0000000000001943. PMID 32483058
- [Background] Day MA, Ehde DM, Burns J, Ward LC, Friedly JL, Thorn BE, Ciol MA, Mendoza E, Chan JF, Battalio S, Borckardt J, Jensen MP. A randomized trial to examine the mechanisms of cognitive, behavioral and mindfulness-based psychosocial treatments for chronic pain: Study protocol. Contemp Clin Trials. 2020 Jun;93:106000. doi: 10.1016/j.cct.2020.106000. Epub 2020 Apr 14. PMID 32302791
- [Background] Day MA, Ciol MA, Mendoza ME, Borckardt J, Ehde DM, Newman AK, Chan JF, Drever SA, Friedly JL, Burns J, Thorn BE, Jensen MP. The effects of telehealth-delivered mindfulness meditation, cognitive therapy, and behavioral activation for chronic low back pain: a randomized clinical trial. BMC Med. 2024 Apr 12;22(1):156. doi: 10.1186/s12916-024-03383-2. PMID 38609994
- [Background] Morone NE, Greco CM, Moore CG, Rollman BL, Lane B, Morrow LA, Glynn NW, Weiner DK. A Mind-Body Program for Older Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):329-37. doi: 10.1001/jamainternmed.2015.8033. PMID 26903081